CLINICAL TRIAL: NCT06862427
Title: A Multi-language Smartphone-based Healthy Lifestyle Intervention for Firefighters: A Cluster Randomized Controlled Trial
Brief Title: A Multi-language Smartphone-based Healthy Lifestyle Intervention for Firefighters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NYCU113176AE; NSTC-111-2314-B-A49A-507-MY3 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Mental Health; Physical Performance; Cardiovascular Health; Lifestyle Intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Healthy Lifestyle APP Intervention (Traditional Chinese Version) (Experimental)
  Interventions: Behavioral: Healthy Lifestyle Application (Traditional Chinese Version)

INTERVENTIONS:
Behavioral: Healthy Lifestyle Application (Traditional Chinese Version) — A firefighter-oriented Healthy Lifestyle Application (Traditional Chinese Version)
  Arms: Healthy Lifestyle APP Intervention (Traditional Chinese Version)

SUMMARY:
The goal of this cluster randomized controlled trial is to evaluate the effects of a smartphone-based Healthy Lifestyle (HLS) intervention on firefighters' mental and physical health in firefighters in Tainan, Taiwan. The main questions it aims to answer are:

* Does the Traditional Chinese version of the HLS mobile App improve firefighters' mental and physical health compared to usual care?
* Can the intervention effectively promote a healthy lifestyle and reduce the risk of chronic non-communicable diseases among firefighters?

Researchers will compare firefighters receiving the smartphone-based HLS intervention to those receiving usual care to determine whether the intervention leads to improved health and fitness outcomes over 3 to 6 months.

Participants will:

* Use the Traditional Chinese version of the HLS mobile App, originally developed at Cambridge Health Alliance, Harvard Medical School, and adapted for firefighters in Taiwan.
* Be randomly assigned to either the intervention group (HLS App) or the control group (usual care).
* Undergo health and fitness assessments at baseline and at 3 to 6 months post-intervention.

Anticipated outcomes are improvements in mental and physical health among firefighters receiving the intervention compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Career firefighters who are older than or equal 20 years old

Exclusion Criteria:

* Career firefighters who are younger than 20 years old
* Firefighters who are retired or are volunteer firefighters.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 3 to 6 months after the intervention starts
  The participants will maintain a quiet sitting posture for at least five minutes, and the measurement will be taken on a healthy arm without any prior surgery or disease. The blood pressure measuring device will be calibrated and will automatically take three measurements, with a one-minute interval between each. The average blood pressure value will be recorded.
Depressive Symptoms | Before the intervention and 3 to 6 months after the intervention starts
  The participants will be asked to complete questionnaires measuring depressive symptoms, which includes the Beck Depression Inventory for Primary Care (BDI-PC) and the Patient Health Questionnaire (PHQ-9). Questions related to self-harm thoughts have been removed from these instruments to eliminate the need for further referrals. Higher scores indicate greater depressive symptoms.
Posttraumatic Stress Disorder Symptoms | Before the intervention and 3 to 6 months after the intervention starts
  The participants will be asked to complete a Posttraumatic Stress Disorder Checklist (PCL-5) questionnaire which measures posttraumatic stress disorder symptoms. Questions related to self-harm thoughts have been removed from these instruments to eliminate the need for further referrals. Higher scores indicate greater depressive symptoms.
Body Mass Index (BMI) | Before the intervention and 3 to 6 months after the intervention starts
  The body mass index (BMI) will be calculated by dividing the weight in kilograms by the square of the height in meters. The height will be self-reported before the intervention and measured to the nearest 0.1 cm while standing upright using a tape measure 3 to 6 months post-intervention, and the weight will be self-reported before the intervention, and measured to the nearest 0.1 kg with a weighing scale 3 to 6 months post-intervention.
Smoking Habit | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will ask if the participants had quit or stopped using tobacco in a questionnaire to verify their smoking habits.
Mediterranean Diet Pattern | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will utilize a Traditional Chinese version of the Mediterranean Diet Score (MDS), consisting of 14 binary questions to determine adherence to the Mediterranean diet pattern.
Overall Physical Activity Levels | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will assess overall physical activity levels over the past 6 months using a Chinese version of a validated physical activity rating (PA-R) questionnaire which our team translated.
Total weekly hours spent sitting | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will ask the participant with the question "Indicate the total number of hours sitting per week"
Average daily hours of sleep | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will ask the participant with the question "Please indicate the total hours of actual sleep in a typical 24-hour period in week"
Frequency of siestas per week | Before the intervention and 3 to 6 months after the intervention starts
  The investigators will ask the participant with the question "How many times do you take a nap per week?"
Glycated Hemoglobin | 3 to 6 months after the intervention starts
  Biochemical parameters will be measured by the cobas b 101 blood testing system (F. Hoffmann-La Roche AG, Basel, Switzerland) with the participants fingertip blood after a 8-hour fasting.
Lipid Profile | 3 to 6 months after the intervention starts
  Biochemical parameters will be measured by the cobas b 101 blood testing system (F. Hoffmann-La Roche AG, Basel, Switzerland) with the participants fingertip blood after a 8-hour fasting.
C-reactive protein(CRP) | 3 to 6 months after the intervention starts
  Biochemical parameters will be measured by the cobas b 101 blood testing system (F. Hoffmann-La Roche AG, Basel, Switzerland) with the participants fingertip blood after a 8-hour fasting.
Physical Performance | In the latter half of 2025
  The participants will provide their semi-annual evaluation reports, including performance metrics in standing long jump, overhead back toss, deadlift, cliffhanger pull-up, 6-meter out-and-back run, farmer's walk, and 1,500-meter run

SECONDARY OUTCOMES:
NT-proBNP | 3 to 6 months after the intervention starts
  Biochemical parameters will be measured by the Cobas h 232 blood testing system (F. Hoffmann-La Roche AG, Basel, Switzerland) with the fingertip blood of participants with hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Fan-Yun Lan Assistant Professor, MD. Ph.D., Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan